CLINICAL TRIAL: NCT04282616
Title: An Exercise Facilitator to Break Down the Barriers to Physical Activity of End-stage Kidney Disease Patients. A Pragmatic Implementation Trial in a Nephrology Unit
Brief Title: An Exercise Facilitator to Activate Simple Training Programs in the Dialysis Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48/2019/Sper/AOUFe
Record Dates: First submitted 2020-02-03; First posted 2020-02-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease Stage 5 on Dialysis
Keywords: exercise; rehabilitation; exercise testing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: End-stage kidney disease patients will be proposed to choose between one of the three organizational models of exercise (counselling; home-based prescription; supervised) or to take part in the project as a control group (no exercise).
Who Masked: Outcomes Assessor
Masking Description: Outcome measures assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Home-based unstructured physical activity program (Experimental): According to each patient's baseline physical activity level, the facilitator will advise patients to start or to increase their spontaneous activity by giving counselling on total exercise time, mode, intensity and frequency as suggested by the American College of Sport Medicine guidelines. Every patient will be provided with a log-book and a wearable physical activity monitor, which has to be returned in the subsequent controls, to favor adherence and objectively measure the exercise activities
  Interventions: Other: Home-based unstructured physical activity program
- Home-based structured low-intensity physical activity program (Experimental): According to each patient's baseline physical activity level, a semi-personalized walking program, will be provided. This program, derived from previous experience on renal patients, includes a 10-min session/day of intermittent walking (1- or 2-min work and 1-min seated rest) to be performed at home at prescribed speed. The speed, converted into walking cadence and followed by a metronome, is weekly increased. Patients will be provided with a daily log containing the detailed exercise prescription and spaces to give a feedback on training execution and related symptoms.
  Interventions: Other: Home-based structured low-intensity physical activity program
- In-hospital structured supervised physical activity program (Experimental): Patients will join the room properly equipped for the exercise program in groups of maximum four subjects for a 2-time/week thirty minutes training sessions, to be performed for dialysis patients immediately before or after the dialysis treatment, or in non-dialysis according to their preferences.
  Each sessions will include low-intensity walking exercises (similar to the structured home-based training), resistance and power exercises with elastic bands and light weights. Each sessions will begin and end with a warm-up and cool-down period of stretching. The total duration of the session will be about 30 minutes. Rate of perceived exertion will be collected and the training intensity will be set according to the patient's baseline capacity and weekly increased.
  Interventions: Other: In-hospital structured supervised physical activity program
- No-training (No Intervention): Patients choosing this option will not start any physical activity program, but they will perform the outcome measures, acting as a control group.

INTERVENTIONS:
Other: Home-based unstructured physical activity program — Counselling on physical activity according to American College of Sports Medicine guidelines
  Arms: Home-based unstructured physical activity program
Other: Home-based structured low-intensity physical activity program — Structured home-based low-intensity intermittent walking program
  Arms: Home-based structured low-intensity physical activity program
Other: In-hospital structured supervised physical activity program — Supervised exercise training program
  Arms: In-hospital structured supervised physical activity program

SUMMARY:
Low physical activity levels and progressive poor functional capacity affect quality of life and clinical outcomes of Chronic Kidney Disease (CKD) patients. Interventions to prevent the functional decline associated with a sedentary lifestyle or to relief from deconditioning are crucial, considering the significant beneficial effects of exercise in all CKD patients, especially in End-stage Kidney Disease patients (ESKD). Unfortunately, physical and psychological barriers to exercise are present and physical activity management is not routinely addressed in the patient's care.

For the first time the project aims to test the impact of the regular presence of an exercise specialist in the Nephrology Unit.

This facilitator, evaluating capacity, motivation and preferences of each patient, will design tailored solutions and assess the related outcomes. Several design of training programs will be proposed to dialysis patients, that can choose the exercise option that best fits their needing.

The study will determine the feasibility of the project, the patients' adherence and the effectiveness of the programs proposed to improve the patients' lifestyle.

DETAILED DESCRIPTION:
The assumption underlying the project is that a wider participation to physical activity programs (PAPs) of ESKD patients may be facilitated by the presence in the Renal Unit of an exercise specialist able to design tailored programs and that this intervention may lead to measurable benefits on physical fitness, quality of life and general health.

The possible different solutions offered by an expert of exercise in chronic diseases might reduce most of the barriers to exercise responsible of the sedentary behavior of the ESKD patients. Aim of the project is to test the impact of the regular presence of this facilitator in a Nephrology Unit in terms of applicability and feasibility as well to identify the preferred and the most effective pathways for the patients.

The identification of a novel cost-effective intervention may represent an important step to manage the change of lifestyle of ESKD patients, to slow down their physical and QoL decline and to reduce hospitalizations and negative outcomes affecting this population.

ELIGIBILITY:
Inclusion Criteria:

* male and females aged > 18 years;
* ability to walk assisted or unassisted at least for 6 meters;
* cognitive functioning to give informed consent identified by a Mini Mental Status Examination score ≥18/30.

Exclusion Criteria:

* severe cardio-respiratory (e.g. unstable angina; severe heart failure identified by New York Heart Association class III or IV);
* neurological or musculoskeletal conditions (e.g. above knee amputation) contraindicating or inhibiting exercise training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
6-minute walking test (Mobility) | Change at 3-month (end of training) respect to baseline
  Subjects will be instructed to walk as far as possible on a 22m walkway in 6 minutes, with their habitual walking device, with the possibility to slow down and rest if necessary. The total distance walked, the pain-free walking distance, and the perceived exertion at the end of the test will be recorded.

SECONDARY OUTCOMES:
10-meter walking test (gait speed) | Change at 3-month (end of training) respect to baseline
  Patients will be positioned at the start of a 10-meter corridor marked with four lines, respectively at 0, 2, 8 and 10 meters from the start. Patients will be asked to walk as fast as they can, but safely, from the first to the last line, using their habitual walking device. A skilled operator will record the time within the two middle lines, that will be converted into speed. Two trails are allowed for this test, and the mean of the two results will be considered
5-time sit-to-stand test (lower limbs strength) | Change at 3-month (end of training) respect to baseline
  This test consists in moving from a sitting position to a standing position on a 42- cm high chair as quick as possible, for five times, with arms folded across the chest. Time will be taken when the test starts, and when the patient lay his/her buttocks on the chair for the fifth time.
Short Form Health Survey (SF-36) (health-related quality of life) | Change at 3-month (end of training) respect to baseline
  This questionnaire consists of 36 items with a score ranging from 0 to 100 divided into 8 domains examining various aspects of health-related QoL. Higher scores correspond to better quality of life.
Short Falls Efficacy Scale (sFES) (fear of falling) | Change at 3-month (end of training) respect to baseline
  This scale is composed of seven 4-point Likert questions about how concerned the patients is about the possibility of falling. The total score ranges from 7 (no concerned about falling) to 28 (highest concern about falling).
Duke Activity Status Index (DASI) (Estimated functional capacity) | Change at 3-month (end of training) respect to baseline
  This is an assessment tool to evaluate the functional capacity of patients through 12 dichotomous (yes/no) questions covering various aspect of life. The total score, ranges from 0 to 58.2 with higher scores that indicate a higher functional capacity.
Beck Depression Inventory - II (BDI-II) | Change at 3-month (end of training) respect to baseline
  This questionnaire, composed of 21 multiple-choice questions, is suitable for measuring the gravity of clinical depression in adults and in diseased populations. The score ranges from 0 (no depression) to 63 (severe depression)
Number and rate of hospitalizations | 6-month and 12-month (follow up)
  Number and rate of all-cause hospitalizations within participants will be collected.
Number and rate of mortality | 6-month and 12-month (follow up)
  Number and rate of all-cause mortality within participants will be collected.
Rate of participation (qualitative outcome) | Baseline
  Rate of patients providing consent compared to the eligible ones will be calculated
Rate of selection of different exercise program proposed (qualitative outcome) | Baseline
  The rate of patients choosing each of the training option proposed will be calculated to determine patients willingness to exercise and patients preferences about training.
Rate of training sessions completed | 3-month (end of program)
  Adherence to the physical activity program chosen will be assessed at the end of the 3-month training period. The total number of training sessions completed in relation to the prescribed ones will be measured by a ratio. The total adherence will range from 0 (0 sessions completed out of 24) to 100% (24 sessions completed out of 24).
6-minute walking test (Mobility) | Change at 6-month (follow-up) respect to baseline
  Subjects will be instructed to walk as far as possible on a 22m walkway in 6 minutes, with their habitual walking device, with the possibility to slow down and rest if necessary. The total distance walked, the pain-free walking distance, and the perceived exertion at the end of the test will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Manfredini, MD, Principal Investigator — University of Ferrara and University Hospital of Ferrara; Alda Storari, MD, Principal Investigator — University Hospital of Ferrara
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published at the end of the trial after deidentification.
  The database of the study will be published in a public repository.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol will be available upon acceptance by a peer-reviewed journal. IPD will be available beginning 6 months following study results publication.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Manfredini F, Lamberti N, Battaglia Y, Straudi S, Belvederi Murri M, Donadi M, Piva G, Fabbian F, Lopez-Soto PJ, Grassi L, Manfredini R, Basaglia N, Storari A. A Personalized Patient-Centered Intervention to Empower through Physical Activity the Patient in the Dialysis Center: Study Protocol for a Pragmatic Nonrandomized Clinical Trial. Methods Protoc. 2020 Dec 6;3(4):83. doi: 10.3390/mps3040083. PMID 33470990